CLINICAL TRIAL: NCT03222154
Title: EFFECTS OF SHOCK WAVE THERAPY IN MIOFASCIAL PAIN: RANDOMIZED AND BLIND CLINICAL TEST
Brief Title: EFFECTS OF SHOCK WAVE THERAPY IN WOMEN WITH PAIN IN TRAPÉZIO MUSCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Marcel Valentim da Silva (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Marcel Valentim da Silva, Principal Investigator, Estácio Ponta Negra
Organization: Estácio Ponta Negra (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFRN
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Pain; Muscle Tonus
Keywords: High Energy Shock Waves; physiotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 3 groups: Control (n = 20), without intervention; Placebo (n = 20), simulation of the application of shock wave therapy; And shock wave therapy (n = 20).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 20 volunteers without intervention. At the end of the study they received an application of shock wave therapy.
- Placebo (Placebo Comparator): 20 volunteers who received simulation of the application of shock wave therapy
  Interventions: Device: Placebo - Shock wave therapy
- Experimental (Experimental): 20 volunteers who received shock wave therapy
  Interventions: Device: Experimental - Shock wave therapy

INTERVENTIONS:
Device: Experimental - Shock wave therapy — Shock wave therapy was performed with the Master Plus 200® Storz Medical equipment, radial emission 2000 pulses, frequency 15 Hz and pressure 1 Bar.
  Other Names: High energy shock wave therapy
  Arms: Experimental
Device: Placebo - Shock wave therapy — Simulation of shock wave therapy
  Arms: Placebo

SUMMARY:
The study consisted of 60 women who had pain-point pains in the upper fibers of the trapezius muscle. They had a medical age of 22.8 years, with a body mass index of 22.8 kg / cm2.They underwent an initial assessment, with a visual analogue pain scale, followed by an assessment of pain threshold, and manual muscle strength.Then, they were allocated into three groups: control group with 20 volunteers without intervention, placebo group with 20 volunteers with shock wave simulation and an intervention group with 20 volunteers with shock wave therapy.

All volunteers were evaluated immediately after the protocol (post evaluation) and 48 hours after the intervention protocol (48 hour evaluation). A mixed ANOVA of repeated measurements was used for intra and intergroup comparisons, followed by tukey post hoc. Significance was set at 5% (p <0.05).

DETAILED DESCRIPTION:
The objective was to investigate the effects of shock wave therapy on the pain of trigger points in the upper fibers of the trapezius muscle.

A randomized, blinded clinical trial of 60 women (mean age 22.8 years and mean body mass index of 22.8 kg / cm2) with presence of trigger points in the upper fibers of the trapezius muscle. These were submitted to an initial evaluation (AV1), composed of the visual analogical pain scale, followed by an evaluation of the pain threshold, using algometry.

Then, the evaluation of the electromyographic activity of the upper trapezius muscle was performed, as well as of its muscular strength by manual dynamometry. Then allocated randomly in 3 groups: Control (n = 20), without intervention; Placebo (n = 20), simulation of the application of shock wave therapy; And shock wave therapy (n = 20).

Shock wave therapy was performed with the Master Plus 200® Storz Medical equipment, radial emission 2000 pulses, 15 Hz frequency and pressure of 1 Bar. All volunteers were evaluated immediately after the protocol (post evaluation) and 48 hours After the intervention protocol (evaluation 48 hours). A mixed ANOVA of repeated measurements was used for intra and intergroup comparisons, followed by tukey post hoc. Significance was set at 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Women with painful symptoms, compatible with the referred pain pattern of trigger points in the upper trapezius muscle.
* Age range of 18 to 35 years.
* No upper limb injury in the last 6 months.
* Featuring trigger points identified in the upper trapezius muscle.
* Present pain and / or moderate and / or severe disability after application of specific instruments.

Exclusion Criteria:

* Present unbearable pain during the evaluation procedures.
* Missing or not executing the solution correctly.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | five minutes
  The subjective pain intensity was evaluated using the Visual Analogue Scale. Which consists of a horizontal line, 10 centimeters long, marked at one end by a rating of 0 - "No Pain" and the other by the classification "Maximum Pain". The patient had to make a line perpendicular to the line, at the point that represents the intensity of his pain.
Evaluation of trigger points | fifteen minutes
  The presence of trigger points was investigated in the upper trapezius muscle on the side that the volunteer reported pain or bilateral.
  The evaluation was performed with the volunteers in the ventral decubitus, and bilaterally evaluated the presence of the trigger points in the upper trapezius. The number of trigger points was recorded according to the classification: active PMG, latent PGM and total PGM. The side that presented a larger number of trigger points was the side used to evaluate the experimental procedures. If the number of active trigger points were equal on both sides, the upper limb considered dominant by the volunteer was chosen for the evaluation.
Evaluation of pressure pain threshold | ten minutes
  To evaluate the pain threshold, a WAGNER® FDM algometer was used, which is a device consisting of a 1 cm2 rubber disc connected to a pressure gauge, which shows values in N.
  The volunteers were previously advised on how the procedure would be performed. And that when when the pressure with the tip of the apparatus began to evoke pain / threshold it was necessary to say loudly the word "Stop"
Electromyographic Evaluation (EMG) Electromyographic Evaluation (EMG) | twenty minutes
  Electromyographic signal processing was performed with a TeleMyo DTS Desk Receiver® electromyography channel (Noraxon USA Inc., Scottsdale, USA) with a 20-500 Hz bandpass filter, gain of 1500 times, and a rejection rate of Common mode greater than 100 dB. The electromyographic evaluation was performed using the bipolar technique, with simple double wireless electrodes.
Strength evaluation | ten minutes
  The muscle strength test was performed with a manual dynamometer (Lafayette® - model 01165), for the force in the shoulder lift movement. For this evaluation the volunteers were seated, with the shoulder in extension position, and consequently the upper limb on the side of the body. The dynamometer was placed in a fixed bulkhead and the shoulder was elevated, resisting the movement and performing an isometric contraction.
Assessment by the Change Perception Scale | ten minutes
  The Patient Global Impression of Change Scale questionnaire was applied in its Portuguese version, Scale of Perception of Change, being an instrument of easy understanding and application. It becomes a useful tool to quantify the perception of change in health status and satisfaction of a treatment of chronic musculoskeletal pain.

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: Starting 6 months after publication